CLINICAL TRIAL: NCT01104701
Title: A Randomized, Multi-dose, Controlled Trial Investigating the Efficacy, Safety and Tolerability, and Pharmacokinetics of Exenatide Once Monthly Suspension.
Brief Title: A Study to Examine the Efficacy, Safety and Tolerability, and Pharmacokinetics of Exenatide Once Monthly Suspension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCB111
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Results first posted 2014-07-17 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-07

CONDITIONS: Type 2 Diabetes
Keywords: Exenatide; Amylin; Lilly; Byetta; Exenatide Once Weekly
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group A (Active Comparator): 2 mg exenatide once weekly subcutaneous (SC). This arm is used as a reference arm in the study.
  Interventions: Drug: exenatide once weekly
- Group B (Experimental): Low dose 5 mg exenatide once monthly suspension SC.
  Interventions: Drug: exenatide once monthly suspension
- Group C (Experimental): Medium dose 8 mg exenatide once monthly suspension SC.
  Interventions: Drug: exenatide once monthly suspension
- Group D (Experimental): High dose 11 mg exenatide once monthly suspension SC.
  Interventions: Drug: exenatide once monthly suspension

INTERVENTIONS:
Drug: exenatide once weekly — subcutaneous injection, 2 mg, once a week
  Arms: Group A
Drug: exenatide once monthly suspension — subcutaneous injection, low dose, once a month
  Arms: Group B
Drug: exenatide once monthly suspension — subcutaneous injection, medium dose, once a month
  Arms: Group C
Drug: exenatide once monthly suspension — subcutaneous injection, high dose, once a month
  Arms: Group D

SUMMARY:
The purpose of Study BCB111 is to collect efficacy, pharmacokinetic, pharmacodynamic, safety, and tolerability data in patients with type 2 diabetes to assess the feasibility of once monthly dosing of the exenatide suspension formulation.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years old at study start
* Has been diagnosed with type 2 diabetes mellitus
* Has HbA1c of 7.1% to 11.0%, inclusive, at study start
* Has been treated with diet and exercise alone or with a stable regimen of metformin, pioglitazone, or a combination of metformin and pioglitazone, for a minimum of 2 months prior to study start
* Either is not treated with or has been on a stable treatment regimen with any of the following medications for a minimum of 2 months prior to study start: hormone replacement therapy (female subjects); antihypertensive agents; thyroid replacement therapy; or antidepressant agents

Exclusion Criteria:

* Clinically significant medical condition that could potentially affect study participation including:
* Acute or chronic pancreatitis
* Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia (MEN) type 2
* Active cardiovascular disease within 3 months of study start
* Underlying hepatic or renal disease
* Inflammatory bowel disease, or other severe gastrointestinal diseases (particularly those that may affect gastric emptying, such as gastroparesis, pyloric stenosis, and metabolic surgery)
* Has had > 2 episodes of major hypoglycemia in the preceding 6 months before study start
* Has received any investigational drug within 30 days (or 5 half-lives of the investigational drug, whichever is greater) prior to study start
* Has been treated, is currently being treated, or is expected to require or undergo treatment with any of the following treatment excluded medications:

  * Any exposure to exenatide (BYETTA®, exenatide once weekly, or exenatide suspension), liraglutide (Victoza®), or any GLP-1 receptor agonist
  * Any DPP-IV inhibitor, sulfonylurea (SU), or rosiglitazone (Avandia®) within 3 months prior to study start
  * Alpha glucosidase inhibitor, meglitinide, nateglinide, or pramlintide (SYMLIN®) within 30 days prior to study start
  * Insulin within 2 weeks prior to study start, or for more than 1 week within 3 months prior to study start
  * Systemic corticosteroids by oral, intravenous, intra-articular, or intramuscular route; or potent, inhaled, or intrapulmonary (including ADVAIR®) steroids known to have a high rate of systemic absorption
  * Prescription or over-the-counter weight loss medications within 3 months prior to study start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2010-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vice President Research and Development, Study Director — Amylin Pharmaceuticals, LLC.
Locations (2):
- United States (2):
  - Research Site, Phoenix, Arizona
  - Research Site, Lincoln, Nebraska

REFERENCES:
- [Derived] Wysham CH, MacConell L, Hardy E. Efficacy and Safety of Multiple Doses of Exenatide Once-Monthly Suspension in Patients With Type 2 Diabetes: A Phase II Randomized Clinical Trial. Diabetes Care. 2016 Oct;39(10):1768-76. doi: 10.2337/dc16-0238. Epub 2016 Jul 19. PMID 27436275

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study initiated 22-May-2010; completed 27-Dec-2010. Once weekly arm: first dose of exenatide administered at study-site on Day 1; self-administered on a weekly basis over subsequent 20 weeks. Once monthly arm: first dose of exenatide administered at study-site on Day 1;self-administered on monthly basis by participants over next 20 weeks.
Groups:
- 2 mg Exenatide Weekly: 2 milligrams (mg) exenatide microspheres in aqueous diluent were administered once a week as a subcutaneous injection (SC) over 20 weeks.
- 5 mg Exenatide Monthly: 5 mg exenatide microspheres in Miglyol 812 were administered once a month SC over 20 weeks. Miglyol is a clear oil mixture of medium chain triglycerides.
- 8 mg Exenatide Monthly: 8 mg exenatide microspheres in Miglyol 812 were administered once a month SC over 20 weeks. Miglyol is a clear oil mixture of medium chain triglycerides.
- 11 mg Exenatide Monthly: 11 mg exenatide microspheres in Miglyol 812 were administered once a month SC over 20 weeks. Miglyol is a clear oil mixture of medium chain triglycerides.
Period: Overall Study
Arm/Group | 2 mg Exenatide Weekly | 5 mg Exenatide Monthly | 8 mg Exenatide Monthly | 11 mg Exenatide Monthly
Started | 30 | 30 | 31 | 30
Completed | 30 | 27 | 29 | 28
Not Completed | 0 | 3 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who were randomized and received at least one dose of study study drug were analyzed in the intent to treat (ITT) population.
Groups:
- 2 mg Exenatide Weekly: 2 milligrams (mg) exenatide microspheres in aqueous diluent were administered once a week as a subcutaneous injection (SC).
- 5 mg Exenatide Monthly: 5 mg exenatide microspheres in Miglyol 812 were administered once a month SC. Miglyol is a clear oil mixture of medium chain triglycerides.
- 8 mg Exenatide Monthly: 8 mg exenatide microspheres in Miglyol 812 were administered once a month SC. Miglyol is a clear oil mixture of medium chain triglycerides. .
- 11 mg Exenatide Monthly: 11 mg exenatide microspheres in Miglyol 812 were administered once a month SC. Miglyol is a clear oil mixture of medium chain triglycerides.
- Total: Total of all reporting groups
Arm/Group | 2 mg Exenatide Weekly | 5 mg Exenatide Monthly | 8 mg Exenatide Monthly | 11 mg Exenatide Monthly | Total
Number analyzed (Participants) | 30 | 30 | 31 | 30 | 121
Age, Customized [Number; unit: participants]
  Less than (<) 65 years of age | 28 | 29 | 26 | 27 | 110
  Greater than, equal to (≥) 65 years of age | 2 | 1 | 5 | 3 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 7 | 13 | 43
  Male | 20 | 17 | 24 | 17 | 78
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 1 | 0 | 2 | 3
  Black or African American | 1 | 4 | 2 | 5 | 12
  White | 28 | 24 | 29 | 23 | 104
  Other | 1 | 1 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 31 | 30 | 121
Mean Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percent of hemoglobin] — HbA1c is measured as a percent (%) of all hemoglobin.
  Percent of hemoglobin | 8.64 (1.19) | 8.54 (1.18) | 8.54 (1.18) | 8.37 (1.34) | 8.52 (1.21)
Category of HbA1c [Number; unit: participants]
  HbA1c < 9.0% | 20 | 18 | 19 | 21 | 78
  HbA1c ≥ 9.0% | 10 | 12 | 12 | 9 | 43

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in HbA1c From Baseline to End of Treatment (Week 20) - Evaluable Population
Description: HbA1c was measured as a percent of total hemoglobin at screening, Baseline, and during treatment on Weeks 4, 8, 12, 16, and 20. Baseline was Day 1, or last measurement prior to first dose of study drug. The Evaluable population was defined as participants who completed study procedures in compliance with the protocol and had adequate exposure to the study drug.
Time Frame: Baseline (Day 1) to 20 weeks
Population: All participants who received at least one dose of study drug, complied with the protocol, had adequate study drug exposure, and had a measurement value on the specified week were included in the analysis of the evaluable population. n=number of participants with measurement value.
Measure: Mean (Standard Error); unit: Percent of Hemoglobin
Groups:
- 8 mg Exenatide Monthly: 8 mg exenatide microspheres in Miglyol 812 were administered once a month SC over 20 weeks. Miglyol is a clear oil mixture of medium chain triglycerides. .
Arm/Group | 2 mg Exenatide Weekly | 5 mg Exenatide Monthly | 8 mg Exenatide Monthly | 11 mg Exenatide Monthly
Number analyzed (Participants) | 29 | 26 | 28 | 27
Percent of Hemoglobin
  Change from baseline at Week 4 (n=29, 26, 28, 27) | -0.52 (0.095) | -0.33 (0.127) | -0.24 (0.139) | -0.34 (0.074)
  Change from baseline at Week 8 (n=25, 22, 25, 27) | -1.15 (0.157) | -0.89 (0.200) | -1.03 (0.218) | -0.91 (0.110)
  Change from baseline at Week 12 (n=29, 26, 28, 27) | -1.43 (0.223) | -1.30 (0.209) | -1.19 (0.246) | -1.26 (0.156)
  Change from baseline at Week 16 (n=29, 26, 28, 27) | -1.58 (0.216) | -1.40 (0.215) | -1.41 (0.271) | -1.43 (0.177)
  Change from baseline at Week 20 (n=29, 26, 28, 27) | -1.54 (0.234) | -1.29 (0.210) | -1.31 (0.313) | -1.45 (0.179)

2. Secondary Outcome: Percentage of Participants Achieving HbA1c Target Values at Week 20 - Evaluable Population
Description: HbA1c was measured as a percent (%) of total hemoglobin. The Target values for HbA1c were <7% and ≤ 6.5% at Week 20. Evaluable population was defined as participants who completed study procedures in compliance with the protocol and had adequate exposure to the study drug.
Time Frame: Week 20
Population: All participants who received at least one dose of study drug, complied with the protocol, had adequate study drug exposure, and had a measurement value for Week 20 were included in the analysis of the evaluable population. n=number of participants with measurement value.
Measure: Number; unit: percentage of Participants
Arm/Group | 2 mg Exenatide Weekly | 5 mg Exenatide Monthly | 8 mg Exenatide Monthly | 11 mg Exenatide Monthly
Number analyzed (Participants) | 29 | 26 | 28 | 27
percentage of Participants
  < 7.0% HbA1c | 48.3 | 50.0 | 57.1 | 70.4
  ≤ 6.5% HbA1c | 44.8 | 26.9 | 39.3 | 48.1

3. Secondary Outcome: Mean Change in Body Weight From Baseline to Week 20 - Evaluable Population
Description: Body weight was measured in kilograms (kg) at Baseline, and during treatment at Weeks 2, 4, 6, 8, 9-11, 12, 13, 14, 15, 16, 17-19, and 20. Baseline was Day 1, or last measurement prior to first dose of study drug. Evaluable population was defined as all participants who completed study procedures in compliance with the protocol and had adequate exposure to the study drug.
Time Frame: Baseline (Day 1) to Week 20
Population: All participants who received at least one dose of study drug, complied with the protocol, had adequate study drug exposure, and had a measurement value on the specified week were included in the analysis. n=number of participants with measurement value.
Measure: Mean (Standard Error); unit: kg
Arm/Group | 2 mg Exenatide Weekly | 5 mg Exenatide Monthly | 8 mg Exenatide Monthly | 11 mg Exenatide Monthly
Number analyzed (Participants) | 29 | 26 | 28 | 27
kg
  Change from baseline to Week 2 (n=29,26,28,27) | -0.31 (0.274) | 0.32 (0.232) | 0.31 (0.234) | 0.35 (0.204)
  Change from baseline to Week 4 (n=29,26,28,27) | -0.66 (0.321) | -0.04 (0.249) | 0.32 (0.299) | 0.03 (0.226)
  Change from baseline to Week 6 (n=29,26,28,27) | -1.26 (0.359) | -0.74 (0.304) | -0.45 (0.409) | -0.74 (0.326)
  Change from baseline to Week 8 (n=28,26,28,27) | -1.36 (0.455) | -0.85 (0.395) | -0.33 (0.482) | -0.70 (0.466)
  Change from baseline to Weeks 9-11 (n=29,26,28,27) | -1.73 (0.565) | -0.57 (0.469) | -0.49 (0.498) | -0.83 (0.563)
  Change from baseline to Week 12 (n=28,26,28,27) | -1.49 (0.573) | -0.91 (0.453) | -0.33 (0.578) | -0.76 (0.502)
  Change from baseline to Week 13 (n=29,26,28,27) | -1.96 (0.505) | -1.20 (0.572) | -0.56 (0.591) | -0.97 (0.551)
  Change from baseline to Week 14 (n=29,26,28,27) | -1.91 (0.643) | -0.96 (0.611) | -0.76 (0.589) | -0.81 (0.563)
  Change from baseline to Week 15 (n=29,26,28,26) | -1.84 (0.511) | -1.34 (0.648) | -0.80 (0.581) | -1.24 (0.581)
  Change from baseline to Week 16 (n=29,26,28,27) | -1.85 (0.590) | -1.33 (0.673) | -0.26 (0.551) | -1.02 (0.574)
  Change from baseline to Weeks 17-19(n=29,26,28,27) | -1.63 (0.592) | -1.17 (0.697) | -0.58 (0.629) | -1.72 (0.700)
  Change from baseline to Week 20 (n=29,26,28,27) | -1.36 (0.641) | -1.10 (0.774) | -0.41 (0.559) | -1.14 (0.676)

4. Secondary Outcome: Mean Change in Fasting Glucose From Baseline to Week 20 - Evaluable Population
Description: Fasting glucose was measured in milligrams per deciliter (mg/dL) at screening, Baseline, and during treatment at Weeks 2, 4, 6, 8, 9-11, 12, 13, 14, 15, 16, 17-19, and 20. Baseline was Day 1, or last measurement prior to first dose of study drug. Evaluable population was defined as all participants who completed study procedures in compliance with the protocol and had adequate exposure to the study drug.
Time Frame: Baseline (Day 1) to Week 20
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | 2 mg Exenatide Weekly | 5 mg Exenatide Monthly | 8 mg Exenatide Monthly | 11 mg Exenatide Monthly
Number analyzed (Participants) | 29 | 26 | 28 | 27
mg/dL
  Change from baseline to Week 2 (n=29, 26, 28,27) | -1.16 (8.54) | -12.9 (7.57) | -14.6 (6.36) | -23.5 (5.17)
  Change from baseline to Week 4 (n=29, 25, 28,27) | -21.7 (7.97) | -18.0 (5.96) | -14.2 (8.57) | -23.1 (7.83)
  Change from baseline to Week 6 (n=28, 26, 28,27) | -32.8 (8.58) | -42.6 (5.72) | -39.5 (9.49) | -48.8 (7.67)
  Change from baseline to Week 8 (n=28, 26, 28,27) | -40.8 (8.70) | -45.7 (6.44) | -36.8 (7.45) | -44.0 (7.24)
  Change from baseline to Weeks 9-11 (n=29,26,27,27) | -32.8 (8.77) | -40.2 (8.25) | -44.3 (7.71) | -48.1 (7.60)
  Change from baseline to Weeks 12 (n=29,26,27,27) | -44.8 (10.28) | -37.4 (8.61) | -45.4 (6.78) | -44.9 (7.53)
  Change from baseline to Weeks 13 (n=29,26,28,27) | -42.0 (8.60) | -38.0 (7.52) | -48.6 (6.21) | -45.7 (8.60)
  Change from baseline to Weeks 14 (n=29,26,28,27) | -36.3 (10.51) | -37.3 (7.75) | -47.5 (7.83) | -51.6 (8.68)
  Change from baseline to Weeks 15 (n=29,26,28,26) | -38.0 (11.09) | -37.3 (7.65) | -46.9 (7.35) | -53.1 (8.96)
  Change from baseline to Weeks 16 (n=29,26,28,27) | -34.5 (9.96) | -31.6 (9.24) | -43.3 (10.14) | -46.3 (7.90)
  Change from baseline to Weeks17-19 (n=29,26,28,27) | -33.3 (8.58) | -42.4 (7.16) | -34.6 (9.32) | -55.1 (8.92)
  Change from baseline to Week 20 (n=29,26,28,27) | -34.2 (8.99) | -25.1 (8.49) | -29.8 (9.88) | -48.9 (9.35)

5. Secondary Outcome: Time Weighted Average Concentration and Peak to Trough of Exenatide From Week 12 Through Week 16 - Pharmacokinetic Evaluable - Steady State Population
Description: All participants received an initial blood draw prior to the first dose and a single blood sample was collected at all other subsequent visits, for plasma exenatide assessments and the characterization of pharmacokinetic (PK) parameters following multiple monthly doses over the study period. Exenatide was measured using a validated enzyme-linked immunosorbent assay (ELISA). Time weighted average concentration (Cave (2016-2688 h) and Peak to Trough were measured in picograms per milliliter (pg/mL).
Time Frame: Day 1 to Week 20
Population: PK Evaluable- Steady-State: from trough to trough following Week 12 through Week 16, 3 or more values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | 2 mg Exenatide Weekly | 5 mg Exenatide Monthly | 8 mg Exenatide Monthly | 11 mg Exenatide Monthly
Number analyzed (Participants) | 25 | 24 | 25 | 23
pg/mL
  Cave(2016-2688h) pg/mL | 262.92 (83.54) | 127.13 (69.34) | 247.38 (81.63) | 218.07 (73.77)
  Peak-Trough (2016-2688h) pg/mL | 171.27 (73.85) | 198.06 (86.76) | 424.47 (70.27) | 328.52 (86.30)

6. Secondary Outcome: Mean Change From Baseline in Diastolic and Systolic Blood Pressure at Week 20 - Intent to Treat (ITT) Population
Description: Baseline was Day 1, or last measurement prior to first dose of study drug. Vital signs were measured after the participant had rested for approximately 5 minutes and with the participant in a sitting position. Measurement was recorded in millimeters of mercury (mmHg). The blood pressure measurement was repeated after at least 30 seconds and the average of the two readings recorded. ITT population was defined as all participants who received at least one dose of the study drug.
Time Frame: Baseline (Day 1), Week 20
Population: Participants who received at least one dose of study drug were analyzed in the Intent to Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 2 mg Exenatide Weekly | 5 mg Exenatide Monthly | 8 mg Exenatide Monthly | 11 mg Exenatide Monthly
Number analyzed (Participants) | 30 | 30 | 31 | 30
mmHg
  Diastolic Blood Pressure | -1.7 (8.55) | 3.4 (8.54) | 1.8 (9.61) | 1.9 (8.17)
  Systolic Blood Pressure | -2.3 (13.64) | 4.4 (18.68) | 0.5 (13.97) | 5.0 (12.04)

7. Secondary Outcome: Mean Change From Baseline in Heart Rate at Week 20 - Intent to Treat (ITT) Population
Description: Baseline was Day 1, or last measurement prior to first dose of study drug. Heart rate was measured after the participant had rested for approximately 5 minutes and with the participant in a sitting position. Measurement was recorded in beats per minute (bpm). The measurement was repeated after at least 30 seconds and the average of the two readings recorded. ITT population was defined as all participants who received at least one dose of the study drug.
Time Frame: Baseline (Day 1), Week 20
Population: Participants who received at least one dose of study drug were analyzed in the ITT population.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | 2 mg Exenatide Weekly | 5 mg Exenatide Monthly | 8 mg Exenatide Monthly | 11 mg Exenatide Monthly
Number analyzed (Participants) | 30 | 30 | 31 | 30
bpm | 2.8 (9.58) | 3.9 (10.69) | 5.6 (10.84) | -0.3 (11.55)

8. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs), Serious AEs (SAEs), and AEs Leading to Discontinuation - ITT Population
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. All participants who received at least one dose of study drug were included in the ITT analysis. Treatment-emergent (TE) adverse events were defined as those with onset at or after initiation of study medication on Day 1 through study termination or early termination.
Time Frame: Day 1 to Study Termination (24 Weeks) or early Termination
Population: All participants who received at least one dose of study drug were included in the ITT analysis.
Measure: Number; unit: participants
Arm/Group | 2 mg Exenatide Weekly | 5 mg Exenatide Monthly | 8 mg Exenatide Monthly | 11 mg Exenatide Monthly
Number analyzed (Participants) | 30 | 30 | 31 | 30
participants
  Treatment-Emergent AES | 27 | 25 | 20 | 24
  Treatment-Emergent SAEs | 0 | 2 | 0 | 0
  Treatment-Emergent AEs Leading to Discontinuation | 0 | 0 | 0 | 1

9. Secondary Outcome: Number of Participants With Injection Site Reaction Treatment Emergent Adverse Events - ITT Population
Description: AE is any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. Injection site related adverse events were defined as the adverse events with 'injection site' phrase in preferred term excluding 'injection site nodule'. The following events were Injection Site Reaction AEs: erythema, hematoma, hemorrhage, site pain, site papule, site pruritus, site warmth.
  Participants receiving study drug monthly received 5 injections with last injection at Week 16; Participants receiving study drug weekly received 20 injections with last injection at Week 19.
  .
Time Frame: Day 1 through study termination (Week 24) or early termination.
Population: All participants who received at least one dose of study drug were analyzed in the ITT population.
Measure: Number; unit: participants
Arm/Group | 2 mg Exenatide Weekly | 5 mg Exenatide Monthly | 8 mg Exenatide Monthly | 11 mg Exenatide Monthly
Number analyzed (Participants) | 30 | 30 | 31 | 30
participants | 6 | 8 | 3 | 6

10. Secondary Outcome: Participants Negative or Positive for Anti-exenatide Antibodies - ITT Population
Description: Serum titers of antibodies to exenatide were evaluated using a validated enzyme-linked immunosorbent assay (Covance Method No. ELISA-0308). Positive antibody to exenatide titer: observed at the indicated visit following a negative or missing titer at baseline, or a positive titer that has increased by at least 3 dilutions at the indicated visit from a detectable baseline. Baseline=Day 1.
Time Frame: Day 1 to Study Termination (24 weeks) or early termination
Population: n=all participants who received at least one dose of study drug and had available titer.
Measure: Number; unit: participants
Arm/Group | 2 mg Exenatide Weekly | 5 mg Exenatide Monthly | 8 mg Exenatide Monthly | 11 mg Exenatide Monthly
Number analyzed (Participants) | 30 | 30 | 30 | 30
participants
  Week 2 Negative (n=30,30,30,30) | 27 | 30 | 30 | 29
  Week 2 Low Titer (<625)(n=30,30,30,30) | 3 | 0 | 0 | 1
  Week 2 High Titer (≥625)(n=30,30,30,30) | 0 | 0 | 0 | 0
  Week 20 Negative (n=30,26,29,28) | 7 | 8 | 9 | 9
  Week 20 Low Titer (<625)(n=30,26,29,28) | 15 | 10 | 15 | 15
  Week 20 High Titer (≥625)(n=30,26,29,28) | 8 | 8 | 5 | 4

11. Secondary Outcome: Number of Hematology Laboratory Values of Potential Clinical Importance Observed During Treatment Period - ITT Population
Description: Potential clinical importance are the following: Hematocrit values for males less than (<) 36%, females < 30%; hemoglobin for males <12 grams per deciliter (g/dL), females < 10 g/dL; low platelet values <75,000/micro liter (µL), high values greater than (>) 500,000 µL. Laboratory samples were obtained at baseline (Day 1 or if unavailable, last measurement prior to first study drug dose), Weeks 6, 12, 20, and at study termination (Week 24) or early termination. Number of laboratory values of potential clinical importance presented for Weeks 6 - Week 24 or early termination.
Time Frame: Day 1 to study termination (24 weeks) or early termination
Population: n= all participants who received at least one dose of study drug and had available laboratory measurements.
Measure: Number; unit: laboratory values
Arm/Group | 2 mg Exenatide Weekly | 5 mg Exenatide Monthly | 8 mg Exenatide Monthly | 11 mg Exenatide Monthly
Number analyzed (Participants) | 30 | 30 | 30 | 30
laboratory values
  Week 6 Hematocrit (n=30,30,30,30) | 0 | 1 | 0 | 0
  Hematocrit at study termination (n=30,27,29,28) | 0 | 1 | 0 | 0
  Week 12 Platelets (n=30, 29, 30, 28) | 0 | 1 | 0 | 0

12. Secondary Outcome: Number of Chemistry Laboratory Values of Potential Clinical Importance Observed During Treatment Period - ITT Population
Description: Potential clinical importance (PCI): triacylglycerol lipase high values were > 3* upper limit of normal (ULN); creatinine high values in males >1.6 mg/dL, females >1.4 mg/dL; gamma glutamyl transferase (GGT) high value >3* ULN; bilirubin high value > 2 mg/dL; Urate high values > 10 (males), >8 (females) mg/dL; potassium low value < 3 milliequivalents per liter (mEq/L), high value >5.5 mEq/L; calcium low value < 8 mg/dL and high value > 11 mg/dL. Laboratory samples were obtained at baseline (Day 1 or if unavailable, last measurement prior to first study drug dose), Weeks 6, 12, 20, and at study termination (Week 24) or early termination. Number of laboratory values of potential clinical importance (values could be either low or high) are presented for Weeks 6 - Week 24 or early termination. Note: those tests with no values meeting the PCI criteria, ie, 0 values observed across all treatment arms, are not presented.
Time Frame: Day 1 to Study Termination (Week24) or early termination
Population: All participants who were randomized and received at least one dose of study drug were analyzed in the intent to treat (ITT) population. n= all participants who received at least one dose of study drug and had available laboratory measurements.
Measure: Number; unit: laboratory values
Arm/Group | 2 mg Exenatide Weekly | 5 mg Exenatide Monthly | 8 mg Exenatide Monthly | 11 mg Exenatide Monthly
Number analyzed (Participants) | 30 | 30 | 31 | 30
laboratory values
  triacylglycerol lipase Week 12 (n=30,29,29,28) | 1 | 1 | 0 | 0
  triacylglycerol lipase Week 20 (n=30,27,29,28) | 1 | 0 | 0 | 1
  Creatinine Week 6 (n=30,30,30,30) | 0 | 1 | 0 | 0
  Creatinine Week 12 (n=30,29,30,28) | 1 | 0 | 0 | 0
  Creatinine Week 20 (n=30,26,28,28) | 0 | 1 | 0 | 0
  Creatinine at study termination (n=30,26,29,28) | 0 | 0 | 1 | 0
  GGT Week 6 (n=30,30,30,30) | 2 | 0 | 0 | 0
  GGT Week 20 (n=30,26,28,28) | 1 | 0 | 1 | 0
  GGT study termination (n=30,26,29,28) | 1 | 0 | 1 | 0
  Bilirubin Week 6 (n=30,30,30,30) | 0 | 1 | 0 | 0
  Bilirubin Week 12 (n=30,29,30,28) | 0 | 1 | 0 | 0
  Urate Week 6 (n=30,30,30,30) | 1 | 1 | 2 | 2
  Urate Week 12 (n=30,29,30,28) | 0 | 3 | 1 | 2
  Urate Week 20 (n=30,26,28,28) | 0 | 1 | 2 | 2
  Urate Study termination (n=30,26,29,28) | 1 | 0 | 0 | 0
  Potassium Week 6 (n=30,30,30,30) | 1 | 0 | 0 | 0
  Calcium Week 6 (n=30,30,30,30) | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 to Week 24 or early termination
Description: Note: Injection site related adverse events were defined as adverse events with 'injection site' phrase in Preferred Term excluding 'injection site nodule'.
Arm/Group | 2 mg Exenatide Weekly | 5 mg Exenatide Monthly | 8 mg Exenatide Monthly | 11 mg Exenatide Monthly
Serious Adverse Events (participants affected / at risk) | 0/30 | 2/30 | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 27/30 | 25/30 | 20/31 | 24/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 mg Exenatide Weekly (N=30) | 5 mg Exenatide Monthly (N=30) | 8 mg Exenatide Monthly (N=31) | 11 mg Exenatide Monthly (N=30)
Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 2 mg Exenatide Weekly (N=30) | 5 mg Exenatide Monthly (N=30) | 8 mg Exenatide Monthly (N=31) | 11 mg Exenatide Monthly (N=30)
Headache (Nervous system disorders) | 9 | 5 | 7 | 8
Nausea (Gastrointestinal disorders) | 4 | 5 | 7 | 7
Diarrhea (Gastrointestinal disorders) | 8 | 2 | 4 | 5
Decreased Appetite (Metabolism and nutrition disorders) | 4 | 1 | 3 | 6
Vomiting (Gastrointestinal disorders) | 3 | 2 | 4 | 5
Injection site pruritus (General disorders) | 5 | 4 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 3 | 1 | 5 | 3
Eructation (Gastrointestinal disorders) | 0 | 2 | 4 | 4
Injection site erythema (General disorders) | 4 | 2 | 1 | 2
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 3 | 1
Fatigue (General disorders) | 1 | 1 | 3 | 3
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 3 | 0 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 3
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Flatulence (Gastrointestinal disorders) | 1 | 1 | 3 | 1
Injection site Hematoma (General disorders) | 2 | 0 | 0 | 1
Injection site hemorrhage (General disorders) | 0 | 1 | 1 | 2
Injection site pain (General disorders) | 1 | 1 | 0 | 2
Pain (General disorders) | 2 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 1 | 1 | 2
Sinusitis (Infections and infestations) | 2 | 1 | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 2 | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 3 | 1
Anxiety (Nervous system disorders) | 0 | 2 | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.